CLINICAL TRIAL: NCT03073031
Title: The Use of PRO-CTCAE by Patients Receiving Immunotherapy for the Treatment of Malignant Melanoma
Brief Title: The Use of PatientReportedOutcomes (PRO)- CTCAE by Melanoma Patients Receiving Immunotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: REHPA, The Danish Knowledge Centre for Rehabilitation and Palliative Care (Other); Rigshospitalet, Denmark (Other); Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Laerke Kjaer Tolstrup, Principal investigator, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SDUSF-2016-90/R1 - (548)
Record Dates: First submitted 2016-10-31; First posted 2017-03-08 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Adverse Effects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Patients report their adverse events on a tablet once a week (intervention) as a supplement to having them monitored every 3 weeks by a physician
  Interventions: Device: Tablet: Samsung Galaxy Tab A
- Control (No Intervention): Patients have their side effects monitored by a physician every 3 weeks (control)

INTERVENTIONS:
Device: Tablet: Samsung Galaxy Tab A
  Arms: Intervention

SUMMARY:
This study evaluates if melanoma patients who report their side effects to immunotherapy weekly by the use of ePRO-CTCAE will experience an overall reduction of grade 3 and 4 events with 50% compared to routine monitoring carried out every 3 weeks.

DETAILED DESCRIPTION:
Hypothesis:

- Melanoma patients who report their side effects to immunotherapy by the use of PRO-CTCAE (Common Terminology Criteria for Adverse Events) will experience an overall reduction of grade 3 and 4 events with 50% compared to routine monitoring.

Aim:

* Primary endpoint: To examine if the electronic tool PRO-CTCAE used on a weekly basis by patients receiving immunotherapy to supplement standard AE monitoring, results in cutting the frequency of grade 3 or 4 adverse events during treatment by 50% compared to patients who get a standard AE monitoring schedule every 3 weeks.
* Secondary endpoints: 1)To examine if the time patients experience grade 2 or higher toxicity, differs in the two groups 2)To examine if more symptoms are reported in the intervention group 3) To examine if there is a difference between the 2 group when it comes to number of extra out-patient visits, days in hospital, telephone consultations and days in prednisone therapy 4) To examine if PRO-CTCAE is implementable in daily practice (will be explored in study 2 and 3).
* Exploratoty endpoint: To examine, using both qualitative and quantitative data, patients´ and clinicians´ experiences with the e-Health intervention to monitor side effects during treatment with immunotherapy in routine clinical practice.

Method:

All patients who are about to receive immunotherapy for the treatment of malignant melanoma at the Department of Oncology, Odense University Hospital (OUH), will be asked to participate. Patients who meet eligibility criteria will be randomized in a 1:1 ratio to either the intervention arm (the use of PRO-CTCAE) or the control arm (standard AE monitoring schedule). Approximately 70 patients in each arm. Inclusion will take place between September 2016 and July 2018. Patients in the intervention arm will report their events weekly for the first 12 weeks of treatment. Clinical staff and patients in the intervention arm will receive instructions on how to use the Ambuflex system to complete the electronic PRO-CTCAE questionnaire (patients) and include the reports in daily practice (clinical staff). Assistance from clinical staff will be provided to patients when needed. Moreover, hospital staff will receive education and written instructions on how to handle the weekly feedback form the patients in the intervention arm.

Evaluation: Studies show that 16% of patients treated with Pembrolizumab/Nivolumab experience grade 3 or 4 side effects during treatment. When it comes to Ipilimumab, the number is 27% and when the drugs are combined the number is as high as 55 %. It is however not all adverse events which the patients can report themselves and when biochemical AEs are deducted, it is estimated that the numbers suitable for self-reporting are as follows: Pembrolizumab/Nivolumab 10%, Ipilimumab 20%, Combination therapy 40%.The primary endpoint of the randomized trial is to reduce the frequency of grade 3 or 4 side effects from 10% to 5% for pembrolizumab /Nivolumab, from 20% to 10 % for Ipilimumab and from 40% to 20% for the combination theory. Realistically, 140 patients can be included in the course of 2 year according to the Danish Melanoma Group. A level of significance of 0.2 is accepted reaching a power of 0.61 for Pembrolizumab/Nivolumab, 0.80 for Ipilimumab) and 0,96 for the combination therapy. These numbers are acceptable due to the fact that this is a pilot study; PRO-CTCAE has not been used in connection with immunotherapy prior to this study and only in a few projects with other patients in Denmark. Moreover, it is prioritized that the Department of Oncology, OUH is the only site, so that the applicant can make sure that all relevant patients are recruited and that clinicians are constantly reminded of the project. Also, the applicant will be able to teach both patients and clinicians on how to use the tool. All in all, the collection of data will be easier and of a higher quality when the study is only being conducted in one site.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years of age
* who read and understand Danish,
* who have been diagnosed with malignant melanoma,
* who are about to be treated with immunotherapy for their disease (1st and 2nd line, mono-therapy and combination therapy).
* Moreover, patients must have signed and dated a written informed consent form in accordance with regulatory and institutional guidelines and 6) be willing and able to comply with the completion of PRO-CTCAE and other required questionnaires.

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
The number of patients who experience drug-related grade 3 or 4 adverse events assessed by CTCAE 4.0 will be reduced by 50% in the intervention arm compared to patients in the control arm | The first 6 months of treatment with immunotherapy

SECONDARY OUTCOMES:
The time patients experience grade 2 or higher toxicity assessed by CTCAE, differs in the intervention arm and the control arm respectively | The first 6 months of treatment with immunotherapy
The number of drug-related adverse events assessed by CTCAE 4.0 reported in the intervention will be higher compared to the adverse events reported in the control arm | The first 6 months of treatment with immunotherapy
The number of contacts to the hospital will be higher in the intervention arm compared to patients in the control arm | The first 6 months of treatment with immunotherapy
The number of hospitalizations are fewer in the intervention arm compared to the control arm. | The first 6 months of treatment with immunotherapy
Patients in the intervention arm receive a lower accumulated prednisone dose compared to patients in the control arm | The first 6 months of treatment with immunotherapy
Patients in the intervention arm have a longer progression free survival compared to patients in the control arm | Estimation of median PFS and progression free survival rate at 6, 12 and 24 months
  PFS is estimated using Kaplan Meier method and differences estimated using logrank test
Patients in the intervention arm have a longer overall survival compared to patients in the control arm | Estimation of median OS and overall survival rate at 6, 12 and 24 months
  OS is estimated using Kaplan Meier method and differences estimated using logrank test
Patients in the intervention arm have a better QoL compared to patients in the control arm | baseline, week 24 and week 48
  EQ-5D-5L and FACT-M questionnaires are used to examine the outcome
The QoL of patients who experience grade 3 or 4 irAEs vs. no grade 3 or 4 irAEs | baseline, week 24 and week 48
  EQ-5D-5L and FACT-M questionnaires are used to examine the outcome

CONTACTS AND LOCATIONS:
Overall Officials: Laerke K. Tolstrup, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tolstrup LK, Pappot H, Bastholt L, Moller S, Dieperink KB. Impact of patient-reported outcomes on symptom monitoring during treatment with checkpoint inhibitors: health-related quality of life among melanoma patients in a randomized controlled trial. J Patient Rep Outcomes. 2022 Jan 21;6(1):8. doi: 10.1186/s41687-022-00414-5. PMID 35061112
- [Derived] Tolstrup LK, Bastholt L, Dieperink KB, Moller S, Zwisler AD, Pappot H. The use of patient-reported outcomes to detect adverse events in metastatic melanoma patients receiving immunotherapy: a randomized controlled pilot trial. J Patient Rep Outcomes. 2020 Oct 30;4(1):88. doi: 10.1186/s41687-020-00255-0. PMID 33125537
- [Derived] Tolstrup LK, Pappot H, Bastholt L, Zwisler AD, Dieperink KB. Patient-Reported Outcomes During Immunotherapy for Metastatic Melanoma: Mixed Methods Study of Patients' and Clinicians' Experiences. J Med Internet Res. 2020 Apr 9;22(4):e14896. doi: 10.2196/14896. PMID 32271150